CLINICAL TRIAL: NCT05420870
Title: A Randomized Controlled Trial to Examine the Effect of Exercise on Bowel Function in Colorectal Cancer Survivors
Brief Title: Effect of Exercise on Bowel Function in Colorectal Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 4-2022-0338
Record Dates: First submitted 2022-05-26; First posted 2022-06-15 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Colorectal Cancer; Low Anterior Resection Syndrome
MeSH Terms: conditions — Colorectal Neoplasms; Low Anterior Resection Syndrome | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental)
  Interventions: Behavioral: exercise
- Usual care group (No Intervention)

INTERVENTIONS:
Behavioral: exercise — Six weeks of exercise intervention
  To meet weekly 150 min of moderate to vigorous physical activity and twice weekly strength exercise General description of the exercise program
  Main goal of the supervised exercise (1 hour per session, twice a week) are three folds. 1) Instruct participants to correctly perform prescribed exercises. 2) Encourage participants to be compliant to exercise program. 3) Participants were encouraged to hand in their exercise diary
  Main goal of the home-based exercise is to perform calisthenics exercise daily. Participants were encouraged to perform at least one set of exercise (8-12 different exercises) and stretching (At least 3 days per week, but preferably most of the days) daily
  Basic 8 exercises which increase ROM and strength of shoulder, lower back, Hip, Knee and ankle Additional 4 exercise to increase core strength and stability
  Arms: Exercise group

SUMMARY:
The survival rate of colorectal cancer patients is increasing due to the development of medical technology. However, many colorectal cancer survivors (CRCs) have bowel dysfunction unlike other cancer survivors. After bowel dysfunction of CRCs was known, many previous studies were conducted to improve bowel dysfunction. Medication, probiotics, Biofeedback training (BFT), Kegel exercise, and sacral nerve stimulation were the methods of intervention research to improve bowel movements in CRCs. Research on randomized control trial of BFT and Kegel exercise is very insufficient. Surgery, chemo, and radiation have a lot of influence on the bowel process of CRCs. In particular, damage to the abdominal muscles, pelvic floor muscles, and autonomic nervous system can also be caused by secondary symptoms such as increased fatigue, reduced physical strength, and musculoskeletal diseases. Therefore, the investigators examine that exercise which can improve fatigue, physical fitness, and musculoskeletal disease affects bowel symptoms of colon cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 19 to 70 who have been diagnosed with Sigmoid colon cancer or rectal cancer have surgery for 6 months or more to less than 3 years
2. Three months after chemo and radiation therapy.
3. Six month after stoma take-down
4. Colorectal cancer patients with a LARS (Low Anterior Reservation Syndrome) questionnaire score of 21 or higher

Exclusion Criteria:

1. Subjects who have problems reading or understanding Korean or who have problems communicating with researchers
2. Subjects who plan to undergo surgery at the same time other than colorectal cancer surgery
3. Metastatic colorectal cancer patients.
4. Subjects who have stoma
5. People who are difficult to exercise in the judgment of the medical staff

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-06-19 (Actual)

PRIMARY OUTCOMES:
Anorectal manometry | Baseline (0 week)
  Anorectal manometry is a test performed to evaluate patients with constipation or fecal incontinence. This test measures the pressures of the anal sphincter muscles, the sensation in the rectum, and the neural reflexes that are needed for normal bowel movements.
Anorectal manometry | endline (7 week)
  Anorectal manometry is a test performed to evaluate patients with constipation or fecal incontinence. This test measures the pressures of the anal sphincter muscles, the sensation in the rectum, and the neural reflexes that are needed for normal bowel movements.

CONTACTS AND LOCATIONS:
Overall Officials: Jae Jun Park, Principal Investigator — Dept. of Internal Medicine, Division of Gastroenterology, Sinchon sevarance Hospital, Younsei university College of Medicine
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No